CLINICAL TRIAL: NCT04777929
Title: The Relationship of Phthalate Exposure During Pregnancy and Preeclampsia
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: SAHoWMU-CR2020-07-210
Record Dates: First submitted 2021-02-28; First posted 2021-03-02 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Phthalate Exposure; Preeclampsia; Estrogen; Progestin
MeSH Terms: conditions — Pre-Eclampsia | interventions — Estrogens; Progesterone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- healthy pregnant woman: pregnant woman without any disease of pregnancy
  Interventions: Other: test Phthalates, estrogen and progesterone
- pregnant woman with preeclampia: pregnant woman with preeclampia but without any other disease of pregnancy
  Interventions: Other: test Phthalates, estrogen and progesterone

INTERVENTIONS:
Other: test Phthalates, estrogen and progesterone — test mothers Phthalates in their urine, and test estrogen and progesterone receptor in placental tissue

SUMMARY:
Phthalates are a group of ubiquitous synthetic endocrine-disrupting chemicals. Fetal and neonatal periods are particularly susceptible to endocrine disorders, which prenatal exposure to phthalates causes. There is increasing evidence concerning the potential endocrine disrupting for phthalate exposure during pregnancy. Prenatal exposure phthalates would disrupt the level of sex hormone in pregnant women, which results in preeclampsia. The relationship of prenatal phthalate exposure with maternal and neonatal outcomes in human beings was often sex-specific associations. Because of the potentially harmful influence of prenatal phthalate exposure, steps should be taken to prevent or reduce phthalate exposure during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Term pregnancy with the gestational age of 37-40 weeks

Exclusion Criteria:

* Maternal systemic diseases (hypertension disorders, immunological diseases) or pregnant complications (polyhydramnios, oligohydramnios, diabetes mellitus, intrahepatic cholestasis of pregnancy)
* Delivery before 37 weeks or after 40 weeks

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Eligible participants is female.
Study Population: The participants include pregnant women meeting the inclusion criteria.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Phthalates in urine | 37 weeks to 40 weeks gestation
  Collect the urine of pregnant women and test the abundance of Phthalates

SECONDARY OUTCOMES:
The female progesterone | 37 weeks to 40 weeks gestation
  Collect the placenta tissue of pregnant women and test the abundance of estrogen progesterone receptor

CONTACTS AND LOCATIONS:
Overall Officials: Ying Hua, Study Director — Second Affiliated Hospital of Wenzhou Medical University
Locations (1):
- department of obstetrics of Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang, China